CLINICAL TRIAL: NCT00577876
Title: Assessment of the Functional Significance of Accessory Pudendal Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-073
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — trimix

ARMS (1):
- 1 (Experimental): Day of Surgery:Patient is admitted through the Preoperative Surgical Center (PSC). If a large APA is identified, then subject will continue on study Dissect APA (without any changes from what is routinely done) with a penile injection of Trimix. Once the initial Doppler Ultrasound is completed, the accessory pudendal artery will be temporarily clamped to stop blood flow. After the artery is clamped, the Doppler Ultrasound will be repeated. We estimate an extension of the surgery no longer than 5 or 10 minutes in comparison to the usual operating time. Once the Doppler Ultrasound is completed, the clamp will be removed and the surgery continued in its usual fashion.
  Interventions: Procedure: Trimix Injection with Doppler Ultrasound

INTERVENTIONS:
Procedure: Trimix Injection with Doppler Ultrasound — In case a large APA was identified, it will be dissected following the usual technique. Upon completion of the dissection, patients will have intracavernosal injection of 10 units (0.1 ml) of a Trimix administered (PGE1 10 mcg/ml, papaverine hydrochloride 30 mg/mL and phentolamine mesylate 1mg/mL.
  Once the patient achieves a pharmacologic erection, the initial Doppler Ultrasound is completed, the accessory pudendal artery will be temporarily clamped to stop blood flow. After the artery is clamped, the Doppler Ultrasound will be repeated. We estimate an extension of the surgery no longer than 5 or 10 minutes in comparison to the usual operating time. Once the Doppler Ultrasound is completed, the clamp will be removed and the surgery continued in its usual fashion.

SUMMARY:
For patients with Prostate Cancer advances in medical technology have enabled us to identify "accessory" (additional) pudendal arteries (called APA) while performing a laparoscopic radical prostatectomy (a scope with a video camera is used during the surgery). APAs running near the prostate gland are identified in approximately 1 in 3 to 4 patients. However, large APAs, like the ones looked for in this study, are identified in 15-18% of all patients. These arteries are preserved more than 80% of the time, depending on their size and location.With this study, we plan to evaluate whether APAs supply blood to the penis and male erections, as well as the amount supplied.

DETAILED DESCRIPTION:
Overall, approximately 50% of patients become impotent (inability to achieve or maintain an erect penis; also called erectile dysfunction) after radical prostatectomy (removal of the prostate). It is already known that postoperative (after surgery) erectile dysfunction does not depend solely on the preservation of the nerves going to the penis, but also to the preservation of the arteries bringing blood to the penis.

Although, the presence and frequency of APAs have been studied, and the ability to preserve them has also been noted, we still do not know how much these arteries contribute to a male's erection. With this study, we plan to evaluate whether APAs supply blood to the penis and male erections, as well as the amount supplied. While there is no immediate benefit to you for participating in the study, these findings will further help our understanding of APA's and the importance in preserving them during surgery.

The primary aim of this study is to determine the proportion of men with APAs for whom APAs contribute to penile blood flow. The secondary aim is to describe peak systolic, diastolic and resistive index velocities of the dorsal artery of the penis before and after clamping of the APA.

ELIGIBILITY:
Inclusion Criteria:

* They have selected a LRP, with or without robotic assistance, by Jonathan Colelman, MD, Bertrand Guillonneau, MD, Vincent Laudone, MD, Raul Parra, MD, or Karim Touijer MD for definitive treatment of their prostate cancer after a full discussion of treatment options.

Exclusion Criteria:

* Patients undergoing Open Radical Prostatectomy
* Patients with prior history of insulin dependent diabetes mellitus
* Patient who have received prior radiation therapy to the pelvis or prostate
* Patients requiring anticoagulation postoperatively
* Known allergy to Phenylephrine, Alprostadil, Papaverine or Phentolamine
* Patients whose systolic blood pressure is below 90 mmHg at the time of evaluation despite routine measures taken by the anesthesiologist at his best criteria.
* Patients with labile hypertension or history of prior priapism
* Patients with penile scarring or penile prosthesis
* Patients with an International Index of Erectile Function score < 24

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of men with APAs for whom APAs contribute to penile blood flow | 18 mo

SECONDARY OUTCOMES:
To describe peak systolic, diastolic and resistive index velocities of the dorsal artery of the penis before and after clamping of the APA. | 18 mo

CONTACTS AND LOCATIONS:
Overall Officials: John Mulhall, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm